CLINICAL TRIAL: NCT05722873
Title: The Effects of Fasting on Reprogramming of Lipid Metabolism and Bone Metabolism
Brief Title: The Metabolic Effects of Intermittent Fasting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pouneh K. Fazeli, MD, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY21120112; R01DK133578 (NIH)
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Normal and Overweight Individuals at High-risk of Diabetes
MeSH Terms: interventions — Body Weight Maintenance; Counseling

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fasting (Experimental): Subjects will fast one-day per week for 12 weeks
  Interventions: Behavioral: Fasting arm
- Fasting with weight maintenance (Experimental): Subjects will fast one-day per week for 12 weeks and maintain body weight
  Interventions: Behavioral: Fasting arm; Behavioral: Weight maintenance
- Counseling (Placebo Comparator): Subjects will be counseled on optimal diet and activity recommendations to maintain/achieve a normal BMI (standard of care)
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Fasting arm — Study participants will fast one day per week for 12 weeks
  Arms: Fasting; Fasting with weight maintenance
Behavioral: Weight maintenance — Study participants will be counseled to maintain body weight
  Arms: Fasting with weight maintenance
Behavioral: Counseling — Study participants will be counseled on optimal diet and activity recommendations for maintaining/achieving a normal BMI
  Arms: Counseling

SUMMARY:
Caloric restriction has beneficial metabolic effects in humans including weight loss and improvement in blood pressure and lipid levels. Intermittent fasting has emerged as a popular alternative to caloric restriction as it does not require daily adherence to a dietary protocol, but whether the benefits of fasting protocols are dependent on weight loss is not known. In this study, the investigators will explore the metabolic effects of fasting and evaluate whether these effects, including negative effects on bone metabolism, are independent of weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ages 21-45 years
2. BMI of at least 21 kg/m2 and up to and including BMI of 29 kg/m2
3. Normal thyroid function
4. Regular menses (women)
5. At least one first-degree relative with type 2 diabetes (T2D) and/or history of gestational diabetes

Exclusion Criteria:

1. Any chronic diseases including hypertension and Type 2 diabetes mellitus
2. Indication for lipid-lowering therapy in non-diabetics, using the more stringent AHA guideline cutoff (LDL>190 or an estimated 10-year ASCVD risk of >7.5%)
3. Chronic medications, including oral contraceptive pills
4. Pregnant and/or breastfeeding
5. History of an eating disorder
6. 25-OH vitamin D level < 20 ng/mL
7. Active substance abuse, including alcohol
8. Subjects with a prior history of intermittent fasting
9. The study physician feels that the subject may not be able to safely complete the protocol or may place themselves at risk by undergoing the protocol

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Triglyceride carbon content and degree of saturation | Baseline, 3 months
  Change in triglyceride carbon content and degree of saturation (% variation explained by both carbon number and double bond number in a regression model) between Baseline and Final Intervention visits
Trabecular bone microarchitecture | Baseline, 3 months
  Change in trabecular bone volume fraction at the radius between Baseline and Final Intervention visits

SECONDARY OUTCOMES:
Insulin sensitivity | Baseline, 3 months
  Change in insulin sensitivity as assessed by hyperinsulinemic-euglycemic clamp between Baseline and Final Intervention visits

CONTACTS AND LOCATIONS:
Overall Officials: Pouneh Fazeli, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified information will be shared upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 12 months after publication. No end date.
Access Criteria: Researchers who wish to access deidentified data.

REFERENCES:
- [Derived] Quaytman JA, David NL, Venugopal S, Amorim T, Beatrice B, Toledo FGS, Miller RG, Steinhauser ML, Fazeli PK. Intermittent fasting for systemic triglyceride metabolic reprogramming (IFAST): Design and methods of a prospective, randomized, controlled trial. Contemp Clin Trials. 2024 Nov;146:107698. doi: 10.1016/j.cct.2024.107698. Epub 2024 Sep 17. PMID 39299543